CLINICAL TRIAL: NCT03555526
Title: Comparison of Genotypic Resistance Guided Versus Susceptibility Testing Guided Therapy for the Third-line Eradication of H. Pylori- a Multicenter Randomized Trial
Brief Title: Genotypic Resistance Guided Therapy for Refractory H. Pylori Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201706037MINC
Record Dates: First submitted 2017-12-14; First posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2017-12

CONDITIONS: H Pylori Infection
MeSH Terms: interventions — Esomeprazole; Amoxicillin; Metronidazole; Levofloxacin; Bismuth; Tetracycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genotypic resistance guided therapy (Experimental): The regimen will be chosen according to the genotyping of 23S rRNA and gyrase A of H. pylori. In the absence of gyrase A mutation, esomeprazole (Nexium), amoxicillin (Amoxicillin), levofloxacin (Cravit), metronidazole (Flagyl) for 14 days will be given. In the presence of gyrase A mutation but in the absence of 23S rRNA mutation, esomeprazole (Nexium), amoxicillin (Amoxicillin), clarithromycin (Klaricid), metronidazole (Flagyl) for 14 days will be given. In the presence of both gyrase A and 23S rRNA mutation, bismuth quadruple therapy including esomeprazole (Nexium), bismuth (KCB), tetracycline, and metronidazole (Flagyl) for 10 days will be given.
  Interventions: Drug: Esomeprazole 40mg; Drug: Amoxicillin; Drug: metronidazole; Drug: Levofloxacin 500mg; Drug: Clarithromycin ER; Drug: Dibismuth trioxide; Drug: tetracycline
- Phenotypic resistance guided therapy (Active Comparator): The regimen will be chosen according to the susceptibility testing result. In the absence of levofloxacin resistance, esomeprazole (Nexium), amoxicillin (Amoxicillin), levofloxacin (Cravit), metronidazole (Flagyl) for 14 days will be given. In the presence of levofloxacin resistance but in the absence of clarithromycin resistance, esomeprazole (Nexium), amoxicillin (Amoxicillin), clarithromycin (Klaricid), metronidazole (Flagyl) for 14 days will be given. In the presence of both levofloxacin and clarithromycin resistance, bismuth quadruple therapy including esomeprazole (Nexium), bismuth (KCB), tetracycline, and metronidazole (Flagyl) for 10 days will be given.
  Interventions: Drug: Esomeprazole 40mg; Drug: Amoxicillin; Drug: metronidazole; Drug: Levofloxacin 500mg; Drug: Clarithromycin ER; Drug: Dibismuth trioxide; Drug: tetracycline

INTERVENTIONS:
Drug: Esomeprazole 40mg — Nexium (esomeprazole), 40mg, bid, for 14 days
  Other Names: Nexium (Sequential)
Drug: Amoxicillin — amoxicillin, 1000mg, bid, for 7 days (day 1-day 7)
  Other Names: Amoxicillin (Sequential)
Drug: metronidazole — metronidazole, 500mg, bid, for 7 days (day 8-14)
  Other Names: Flagyl (sequential)
Drug: Levofloxacin 500mg — levofloxacin 250mg, bid, for 7 days (day 8-14)
  Other Names: Cravit (sequential)
Drug: Clarithromycin ER — clarithromycin 500mg, bid, for 7 days (day 8-14)
  Other Names: Klaricid ER 500 (sequential)
Drug: Esomeprazole 40mg — Nexium (esomeprazole), 40mg, bid, for 10 days
  Other Names: Nexium (bismuth quadruple therapy)
Drug: Dibismuth trioxide — Dibismuth trioxide，KCB F.C. TABLETS，300mg，qid, for 10 days
  Other Names: KCB F.C.; bismuth
Drug: metronidazole — metronidazole, 500mg, tid, for 10 days (day 1-10)
  Other Names: Flagyl (bismuth quadruple)
Drug: tetracycline — tetracycline 500mg, qid, for 10 days
  Other Names: tetracycline (bismuth quadruple therapy)

SUMMARY:
The inviestigators aimed to compare the efficacy of genotypic resistance guided versus susceptibility testing guided therapy in the third line treatment for refractory H. pylori infection.

Hypothesis:The investigators hypothesized that genotypic resistance guided sequential therapy is non-inferior to empiric therapy in the third line treatment for refractory H. pylori infection.

Methods: This multicenter, open label, parallel group, randomized trial will be conducted since 2017.07.20. Adult (≥20 years old) patients who failed from at least two eradication therapies for H. pylori infection will be enrolled. Genotypic and phenotypic resistances will be determined in patients who failed from at least two eradication therapies by polymerase-chain-reaction with direct sequencing and E-test and agar dilution test, respectively. Eligible patients will be randomized into either one of the treatment groups (A) genotypic resistance guided therapy; or (B) susceptibility testing guided therapy.

Outcome Measurement The primary outcome is the eradication rate in the third line treatment (genotypic versus susceptibility testing guided therapy) according to intention-to-treat (ITT) analysis.

DETAILED DESCRIPTION:
The inviestigators aimed to compare the efficacy of genotypic resistance guided versus susceptibility testing guided therapy in the third line treatment for refractory H. pylori infection.

Hypothesis:The investigators hypothesized that genotypic resistance guided sequential therapy is non-inferior to empiric therapy in the third line treatment for refractory H. pylori infection.

Methods: This multicenter, open label, parallel group, randomized trial will be conducted since 2017.07.20. Adult (≥20 years old) patients who failed from at least two eradication therapies for H. pylori infection will be enrolled. Genotypic and phenotypic resistances will be determined in patients who failed from at least two eradication therapies by polymerase-chain-reaction with direct sequencing and E-test and agar dilution test, respectively. Eligible patients will be randomized into either one of the treatment groups (A) genotypic resistance guided therapy; or (B) susceptibility testing guided therapy. Eradication status will be determined by 13C-urea breath test at least 6 weeks after eradication therapy. The stool samples will be collected before, and 2 and 8 weeks and 1 year after eradication therapy to analyze the changes in the antibiotic resistance and microbiota of gut flora. The body weight, waist and hip circumference and serum lipid profile, sugar, and HbA1C levels will also be collected before and 2 weeks, 8 weeks and 1 year after eradication therapy.

Outcome Measurement The primary outcome is the eradication rate in the third line treatment (genotypic versus susceptibility testing guided therapy) according to intention-to-treat (ITT) analysis.

Secondary End Points: the eradication rate according per protocol analysis and the adverse effects

Secondary End Point:

(A) Eradication rate according to per protocol analysis (PP analysis) (B) Frequency of adverse effects (C) The changes in the gut microbiota, antibiotic resistance of the Enterobacteriae, metabolic parameters before and after H. pylori eradication (D) The long term eradication rate and reinfection rate

ELIGIBILITY:
Inclusion Criteria:

* H pylori infection failed after at least two eradication therapies
* aged 20 years or greater
* willingness to receive rescue therapy

Exclusion Criteria:

* aged less than 20 years
* history of gastric resection surgery
* history of allergy to study drugs
* pregnancy or lactating women
* severe underlying illness, such as end stage renal disease, decompensated liver cirrhosis, or non-curative malignancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Eradication rate by intention to treat analysis | 8 weeks

SECONDARY OUTCOMES:
Eradication rate by per protocol analysis | 8 weeks
frequency of adverse effects during eradication therapy | 2 weeks
changes of fecal microbiota | 1 year
  changes of fecal microbiota before and after erdication therapy
reinfection rate | 1 year
  reinfection rate 1 year after eradication therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Ming Liou, MD, PhD, Principal Investigator — National Taiwan University Hospital (recruiting); Yen-Nien Chen, MD, Principal Investigator — National Taiwan University Hospital Hsin-Chu Branch; Yu Jen Fang, MD, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch
Locations (1):
- Jyh-Ming Liou, Taipei, Taiwan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen MJ, Chen PY, Fang YJ, Bair MJ, Chen CC, Chen CC, Yang TH, Lee JY, Yu CC, Kuo CC, Chiu MC, Chou CK, Chen CY, Hu WH, Tsai MH, Hsu YC, Shun CT, Luo JC, Lin JT, El-Omar EM, Wu MS, Liou JM; Taiwan Gastrointestinal Disease and Helicobacter Consortium. Molecular testing-guided therapy versus susceptibility testing-guided therapy in first-line and third-line Helicobacter pylori eradication: two multicentre, open-label, randomised controlled, non-inferiority trials. Lancet Gastroenterol Hepatol. 2023 Jul;8(7):623-634. doi: 10.1016/S2468-1253(23)00097-3. Epub 2023 May 10. PMID 37178702